CLINICAL TRIAL: NCT01987661
Title: German: Einfluss Von Airtrapping Auf Atmung Und Schlaf Bei Nichtinvasiver Beatmung (NIV) Von COPD Patienten
Brief Title: The Effects of Airtrapping on Sleep and Breathing in Non Invasive Ventilation (NIV) in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut für Pneumologie Hagen Ambrock eV (Industry)
Collaborators: Weinmann Geräte für Medizin GmbH + Co. KG (Industry)
Responsible Party: Principal Investigator, Georg Nilius, Head of Helios Klinik Hagen Ambrock, Klinik für Pneumologie, Institut für Pneumologie Hagen Ambrock eV
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Airtrap2013
Record Dates: First submitted 2013-11-13; First posted 2013-11-19 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: COPD; Hypercapnic Respiratory Failure
Keywords: COPD; NIV; Airtrapping; Ventimotion2
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- bilevel ventilation BIPAP ST (Active Comparator): one night, BIPAP ST ventilation with individually optimised pressure parameters and supplemental oxygen if necessary.
  Interventions: Device: BIPAP ST
- BIPAP ST plus Airtrap (Experimental): one night, BIPAP ST ventilation with "Airtrap control", same pressure parameters and oxygen.
  Interventions: Device: BIPAP ST; Device: Airtrap

INTERVENTIONS:
Device: BIPAP ST — non invasive ventilation, individually titrated for each patient, if necessary combined with oxygen, to improve hypercapnic respiratory failure.
  Other Names: Ventimotion 2
Device: Airtrap — Addional to the individally titrated BiPAP ventilation parameters the function "AirTrap Control" is added.
  AirTrap Control helps to prevent dynamic hyperinflation and makes it possible for VENTImotion 2 to automatically regulate to the best frequency and expiration time.
  Other Names: Ventimotion 2, Weinmann
  Arms: BIPAP ST plus Airtrap

SUMMARY:
15 COPD patients will be surveyed in this prospective randomized crossover pilot study concerning non invasive ventilation. Patients will be treated over 2 nights in randomized order with Ventimotion2 (Weinmann) with and without Airtrap Control under Polysomnography (PSG) surveillance including transcutaneous pCO2 measurement. The sleep quality is judged by evaluating the PSG and pCO2 values over night.

Target parameters are respiratory rate, sleep quality and influence of Airtrap Control on pCO2 values over night.

ELIGIBILITY:
Inclusion Criteria:

* Stable respiratory situation
* Clinically required NIV
* Capable of giving consent

Exclusion Criteria:

* Invasive ventilation
* Any other severe physical disease that requires immediate medical assistance
* Acute hypercapnic decompensation with pH <7.30 in routine BGA
* Circumstances that doesn't allow mask ventilation (e.g. facial deformation)
* Participation in a clinical trial within the last 4 weeks
* Pregnancy or nursing period
* Drug addiction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-10; Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
breathing frequency | 2 nights
  breathing frequency measured with the flow signal of a polysomnography during non invasive ventilation over night

SECONDARY OUTCOMES:
mean pCO2 level | 2 nights
  mean pCO2 level over night measured with a transcutanous pCO2 monitor (TOSCA)

OTHER OUTCOMES:
Sleep efficiency | 2 nights
  Sleep efficiency is defined by the relation of "time in bed" to "total sleep time" in the overnight polysomnography protocol

CONTACTS AND LOCATIONS:
Overall Officials: Georg Nilius, MD, Principal Investigator — Helios Klinik Hagen
Locations (1):
- Helios Klinik Hagen, Hagen, North Rhine-Westphalia, Germany